CLINICAL TRIAL: NCT07027085
Title: Investigation of the Effects of Virtual Reality Applications on Sensory Processing, Cognitive Skills, Social Functioning and Disease Symptoms in Individuals Diagnosed With Schizophrenia
Brief Title: Investigation of the Effects of Virtual Reality Applications on Individuals Diagnosed With Schizophrenia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Fatıma Zehra Turan, Lecturer, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NiğdeOHU.OT.
Record Dates: First submitted 2025-06-02; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia Disorders
Keywords: virtual reality; social skill training; cognition; sensory processing
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Device: virtual reality
- control group (No Intervention)

INTERVENTIONS:
Device: virtual reality — The intervention group will be applied 14 sessions of virtual reality application, each session lasting 30 minutes and 2 sessions per week. The sessions will be held in a room allocated for this study in the community mental health center. The device on which the application will be made was determined as Meta Quest 3. The contents to be used in the device were determined to be in line with the areas to be examined.
  Arms: intervention group

SUMMARY:
Despite all the positive facts about the use of virtual reality technology in the assessment and treatment of schizophrenia, there are few publications per year. There are few controlled studies covering the effectiveness of virtual reality programs in the training of cognitive and social skills. In future research, more randomized studies with more robust samples are expected, because the results of experimental studies so far encourage this new treatment approach. Therefore, the aim of this study is to examine the effects of virtual reality application on sensory, social and cognitive areas in individuals with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic disease that can cause serious disability and negatively affect quality of life and functionality. According to the results of studies conducted to date, it is assumed that schizophrenia is a syndrome rather than a single disease due to its different clinical types, clinical appearance, course and treatment responses that vary from patient to patient. Schizophrenia is one of the diseases that cause the most disability worldwide. According to World Health Organization data, schizophrenia is in the top ten list of diseases that cause disability for individuals aged 15-44. Individuals diagnosed with schizophrenia usually experience difficulties in the areas of Sensory Processing, Cognitive Functions and Social Skills. Sensory processing disorders in individuals with schizophrenia affect the processes of perceiving and interpreting environmental stimuli: Sounds, lights or tactile stimuli that are considered ordinary in daily life may become disturbing or there may be difficulty in combining visual and auditory information in a harmonious way. This situation also negatively affects social interactions. For example, Javitt and Freedman stated that sensory processing disorders in schizophrenia are related to both cognitive and social functioning dimensions of the disease.

Social skills are one of the most frequently affected areas in schizophrenia and various impairments can be observed. Difficulty in social interactions, introversion and communication problems are frequently observed. Difficulty in understanding facial expressions, body language or tone of voice, decreased ability to understand the emotional states of others or avoidance of social interactions and isolation can be observed. Pinkham et al. stated that social cognition is a significant problem in schizophrenia and that this situation has a direct effect on social functioning. Individuals with schizophrenia also experience impairments in their ability to recognize and express emotions. Kohler et al. emphasized that emotional processing disorders in schizophrenia make social relationships even more difficult.

Schizophrenia can lead to significant impairments especially in cognitive areas and this can significantly affect the individual's daily life. For example; difficulty in focusing on a sustained task, deficiencies in the ability to retain and use instant information, or impairments in higher-level cognitive functions such as problem solving, planning, and decision making. A meta-analysis found that individuals with schizophrenia had significant disadvantages compared to healthy individuals in all cognitive areas. One study showed that parietal lobe functions (related to motor planning) may be impaired in individuals with schizophrenia and that this situation has effects on motor control. These problems reduce the quality of life of individuals with schizophrenia and make it difficult for them to reintegrate into society. Innovative approaches such as virtual reality offer promising solutions for rehabilitation in these areas.

Virtual reality (VR) is a technology in which users experience the feeling of being in three-dimensional environments created by computers. This technology abstracts the user from the physical world and includes them in a virtual world through special headsets and sensors.

Virtual reality technology is used in various fields today. In recent years, it has been increasingly used in medicine and psychology. It is especially effective as a rehabilitation and treatment tool in various disease groups. Virtual reality applications have various advantages and limitations. Advantages: Individuals receive therapy in a controlled environment, away from the risks they may encounter in the real world. Virtual reality environments offer more realistic and impressive experiences than traditional therapies. Applications can be customized according to the needs of individuals. Virtual reality devices objectively measure and record the individual's behaviors and reactions. Limitations: The cost of virtual reality equipment and access to technology may be limited. Some individuals may experience side effects such as dizziness or nausea in virtual environments. More research is needed on the long-term effectiveness of some applications. Virtual reality applications in schizophrenia are drawing attention as an innovative approach to improving individuals' cognitive, social and sensory functions. Such applications provide an effective alternative to traditional methods by allowing therapeutic interventions in a safe environment. Virtual reality targets several areas where individuals with schizophrenia have difficulties. These include; Social Skills: Provides safe practice of social interactions by simulating real-life social situations.

Sensory Processing and Sensitivity: Sensory tolerance is developed by exposure to environmental stimuli.

Cognitive Rehabilitation: Provides tasks that improve attention, memory, and executive functions.

Delusion and Hallucination Management: Therapies that strengthen the perception of reality are applied.

The available data on virtual reality applications are currently limited due to the small number of studies conducted on the subject, and more research is needed to better evaluate its effectiveness as a treatment. However, current evidence reveals its effectiveness and versatility in successfully treating a variety of psychotic symptoms, including delusions, hallucinations, or cognitive and social skills, and suggests virtual reality as a promising new branch of research and therapy. The existing literature agrees on the safety, tolerability, and long-term durability of the therapeutic effects achieved with virtual reality. Studies have reported a decrease in social anxiety and an increase in self-confidence.

For example, in a randomized controlled trial by Park et al. on the use of virtual reality in the treatment of social skills, it was reported that it showed significant improvements in speaking skills and also provided greater motivation for treatment. Freeman et al. developed a virtual reality application that allowed the individual to reframe these thoughts by interacting with an avatar associated with the content of the delusion. In another study, virtual reality application was found to be effective in reducing the intensity and distress of delusions. Effective results were obtained in virtual reality applications used to improve cognitive functions. La Paglia et al. conducted virtual reality training for cognitive rehabilitation targeting attention and executive functions in patients with schizophrenia. Rus-Calafell et al. suggested that virtual reality intervention could be applied to cognitive rehabilitation, social skills training interventions and virtual reality-assisted therapies for psychosis, could provide a valuable method for assessing the presence of symptoms and has the potential to facilitate learning new emotional and behavioral responses.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with schizophrenia
* Volunteering to participate in the study
* Being an adult between the ages of 18-65
* Not in an acute or exacerbated phase
* Scoring 19 or more on the Mini Mental State Examination

Exclusion Criteria:

* Patients who have another psychological or neurological disease other than schizophrenia
* Who are unable to give their own consent will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination | at the beginning (baseline) and end of the intervention (7 weeks)
  The Mini Mental State Examination was first published by Folstein et al. (1975). It consists of eleven items grouped under five main headings: orientation, recording memory, attention and calculation, recall, and language, and is evaluated out of a total of 30 points.
Social Functioning Assessment Scale | at the beginning (baseline) and end of the intervention (7 weeks)
  The Social Functioning Assessment Scale (SAF) will be used for social functioning. This scale, developed in Turkey, assesses social functioning in schizophrenia patients with 19 items and four sub-dimensions. The factors include interpersonal relationships and entertainment with seven items, self-care with seven items, independent living skills with four items, and work life with one item. The score that can be obtained from the scale is between 19 and 57, with a high score indicating a high level of social functioning.
Adolescent/Adult Sensory Profile | at the beginning (baseline) and end of the intervention (7 weeks)
  The Adolescent/Adult Sensory Profile will be used to examine sensory areas. Adolescent/Adult. Sensory Profile is a scale consisting of 60 items. It evaluates the response of 6 sensory patterns to different sensory stimuli. It is used in adolescents and adults aged 11 and above. The 60 items in the Sensory Profile are divided into four categories, each with 15 items equally divided into four categories, each belonging to a different sensory processing pattern. These are: low registration, sensory seeking, sensory sensitivity, sensory avoidance. Using a five-point Likert scale, participants are asked to rate how often they respond to the sensory event/experience described in each item. Each category results in a score range of 5 to 75. Each age group (11-18, 18-65, and 65 and above) has different norm values. The higher the score, the more characteristics the individual exhibits for sensory processing patterns. For example, the higher the score an individual obtains in the "low-recordin
Schizophrenia Cognitive Assessment Scale | at the beginning (baseline) and end of the intervention (7 weeks)
  The Schizophrenia Cognitive Assessment Scale (SCAS) will be used for cognitive assessment. The Schizophrenia Cognitive Assessment Scale was developed by Keefe and colleagues in 2005 and consists of 20 items to determine the degree of cognitive impairment and its effects on daily functioning in schizophrenia patients. The items included in the scale were developed to evaluate attention, memory, reasoning and problem solving, working memory, language production and motor skills, which are frequently affected by neurocognitive impairment in schizophrenia patients and closely related to psychosocial functioning. The average application time of the scale is 12 minutes. Each of the 20 items is evaluated on a severity level ranging from 1 to 4, with higher scores indicating a greater degree of impairment. Information is obtained from three separate sources: the patient himself/herself, the patient's relative who provides information, and the interviewer, who is the physician who follows the

SECONDARY OUTCOMES:
Scale for the Assessment of Positive Symptoms | at the beginning (baseline) and end of the intervention (7 weeks)
  Scale for the Assessment of Positive Symptoms (SAPS) evaluates the level, distribution and severity of positive symptoms in patients with schizophrenia. It was developed by Andreasen. The reliability of the Turkish form was established by Erkoç et al. It is a six-point Likert-type scale with 4 subscales and 34 items, evaluated by the interviewer. The subscales are hallucinations, delusions, strange behavior and formal thought disorder. The scoring of each item ranges from 0 to 5. The total subscale scores are obtained by adding the subscale items and the total scale score is obtained by adding the subscale total scores. The total score ranges from 0 to 170.
Scale for the Assessment of Negative Symptoms | at the beginning (baseline) and end of the intervention (7 weeks)
  Scale for the Assessment of Negative Symptoms (SANS) evaluates the level, distribution and severity of negative symptoms in patients with schizophrenia. It was developed by Andreasan. The reliability of the Turkish form was established by Erkoç et al. It is a six-point Likert-type measurement scale with 5 subscales and 25 items that is evaluated by the interviewer. The subscales are affective blunting, alogia, apathy, anhedonia and attention deficit. The scoring of each item varies between 0-5 and 25. The total subscale scores are obtained by adding the subscale items. The total scale score is obtained by adding the total subscale scores. The total score varies between 0-125.

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Ömer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erkoç Ş, Arkonaç O, Ataklı C, Özmen E. Negatif semptomları değerlendirme ölçeğinin güvenilirliği ve geçerliliği. Düşünen Adam. 1991;4(2):14-5.
- [Background] Erkoç Ş, Arkonaç O, Ataklı C, Özmen E. Pozitif semptomları değerlendirme ölçeğinin güvenilirliği ve geçerliliği. Düşünen Adam. 1991;4(2):20-4.
- [Background] KİRAS F, İNCEDERE A, ESEN D, GÜRCAN MB, ABUT B, İPÇİ K, et al. Şizofreni Hastaları için Toplumsal İşlevselliği Değerlendirme Ölçeğinin geliştirilmesi: Geçerlilik ve güvenirlik çalışması. Anatolian Journal of Psychiatry/Anadolu Psikiyatri Dergisi. 2018;19.
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Özak N. Şizofreni Hastalarinda Bilişsel Bozukluk Düzeyini Değerlendiren Şizofreni Bilişsel Değerlendirme Ölçeğinin Türkçe Geçerlilik ve Güvenilirlik Çalişmasi: Dokuz Eylul Universitesi (Turkey); 2019.
- [Background] Aydın MŞ. Adolesan/Yetişkin Duyu Profili anketi türkçe uyarlamasının geçerlilik güvenilirlik çalışması. 2015.
- [Background] Rus-Calafell M, Garety P, Sason E, Craig TJK, Valmaggia LR. Virtual reality in the assessment and treatment of psychosis: a systematic review of its utility, acceptability and effectiveness. Psychol Med. 2018 Feb;48(3):362-391. doi: 10.1017/S0033291717001945. Epub 2017 Jul 24. PMID 28735593
- [Background] La Paglia F, La Cascia C, Rizzo R, Sanna M, Cangialosi F, Sideli L, et al. Virtual Reality environments to rehabilitation attention deficits in schizophrenic patients. Annual Review of CyberTherapy and Telemedicine. 2016.
- [Background] Craig TK, Rus-Calafell M, Ward T, Leff JP, Huckvale M, Howarth E, Emsley R, Garety PA. AVATAR therapy for auditory verbal hallucinations in people with psychosis: a single-blind, randomised controlled trial. Lancet Psychiatry. 2018 Jan;5(1):31-40. doi: 10.1016/S2215-0366(17)30427-3. Epub 2017 Nov 23. PMID 29175276
- [Background] Freeman D, Bradley J, Antley A, Bourke E, DeWeever N, Evans N, Cernis E, Sheaves B, Waite F, Dunn G, Slater M, Clark DM. Virtual reality in the treatment of persecutory delusions: randomised controlled experimental study testing how to reduce delusional conviction. Br J Psychiatry. 2016 Jul;209(1):62-7. doi: 10.1192/bjp.bp.115.176438. Epub 2016 May 5. PMID 27151071
- [Background] Park MJ, Kim DJ, Lee U, Na EJ, Jeon HJ. A Literature Overview of Virtual Reality (VR) in Treatment of Psychiatric Disorders: Recent Advances and Limitations. Front Psychiatry. 2019 Jul 19;10:505. doi: 10.3389/fpsyt.2019.00505. eCollection 2019. PMID 31379623
- [Background] Macedo M, Marques A, Queirós C. Virtual reality in assessment and treatment of schizophrenia: a systematic review. Jornal brasileiro de psiquiatria. 2015;64(1):70-81.
- [Background] Bisso E, Signorelli MS, Milazzo M, Maglia M, Polosa R, Aguglia E, Caponnetto P. Immersive Virtual Reality Applications in Schizophrenia Spectrum Therapy: A Systematic Review. Int J Environ Res Public Health. 2020 Aug 22;17(17):6111. doi: 10.3390/ijerph17176111. PMID 32842579
- [Background] Freeman D. Studying and treating schizophrenia using virtual reality: a new paradigm. Schizophr Bull. 2008 Jul;34(4):605-10. doi: 10.1093/schbul/sbn020. Epub 2008 Mar 28. PMID 18375568
- [Background] Ertürk NB, Değirmenci FN. SANAL GERÇEKLİK (VR) TEKNOLOJİLERİNİN MİMARLIK SEKTÖRÜNDEKİ YERİ. Karesi Journal of Architecture.2(2):24-36.
- [Background] Bachofner H, Scherer KA, Vanbellingen T, Bohlhalter S, Stegmayer K, Walther S. Validation of the Apraxia Screen TULIA (AST) in Schizophrenia. Neuropsychobiology. 2022;81(4):311-321. doi: 10.1159/000523778. Epub 2022 Apr 1. PMID 35367989
- [Background] Nuechterlein KH, Barch DM, Gold JM, Goldberg TE, Green MF, Heaton RK. Identification of separable cognitive factors in schizophrenia. Schizophr Res. 2004 Dec 15;72(1):29-39. doi: 10.1016/j.schres.2004.09.007. PMID 15531405
- [Background] Mesholam-Gately RI, Giuliano AJ, Goff KP, Faraone SV, Seidman LJ. Neurocognition in first-episode schizophrenia: a meta-analytic review. Neuropsychology. 2009 May;23(3):315-36. doi: 10.1037/a0014708. PMID 19413446
- [Background] La Paglia F, La Cascia C, Rizzo R, Sideli L, Francomano A, La Barbera D. Cognitive rehabilitation of schizophrenia through NeuroVr training. Stud Health Technol Inform. 2013;191:158-62. PMID 23792865
- [Background] Kohler CG, Walker JB, Martin EA, Healey KM, Moberg PJ. Facial emotion perception in schizophrenia: a meta-analytic review. Schizophr Bull. 2010 Sep;36(5):1009-19. doi: 10.1093/schbul/sbn192. Epub 2009 Mar 27. PMID 19329561
- [Background] Pinkham AE, Penn DL, Green MF, Buck B, Healey K, Harvey PD. The social cognition psychometric evaluation study: results of the expert survey and RAND panel. Schizophr Bull. 2014 Jul;40(4):813-23. doi: 10.1093/schbul/sbt081. Epub 2013 May 31. PMID 23728248
- [Background] Javitt DC, Freedman R. Sensory processing dysfunction in the personal experience and neuronal machinery of schizophrenia. Am J Psychiatry. 2015 Jan;172(1):17-31. doi: 10.1176/appi.ajp.2014.13121691. Epub 2014 Nov 17. PMID 25553496
- [Background] Summakoğlu D, Ertuğrul B. Şizofreni ve tedavisi. Lectio Scientific. 2018;2(1):43-61.
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Uyan TT, Köroğlu A, Hocaoglu C. Şizofreni: Etiyoloji, tanı ve tedavi yaklaşımlarında güncel durum. ERÜ Sağlık Bilimleri Fakültesi Dergisi.10(1):19-35.
- [Background] Jauhar S, Johnstone M, McKenna PJ. Schizophrenia. Lancet. 2022 Jan 29;399(10323):473-486. doi: 10.1016/S0140-6736(21)01730-X. PMID 35093231